CLINICAL TRIAL: NCT02325700
Title: Total Laparoscopic Versus Open Aortic Surgery for Abdominal Aortic Disease. A Prospective Study With Propensity Analysis
Brief Title: Total Laparoscopic Versus Open Aortic Surgery for Abdominal Aortic Disease
Status: Completed | Type: Observational
Sponsor: University of Poitiers (Other)
Responsible Party: Sponsor
Other Study IDs: JBR02
Record Dates: First submitted 2014-12-21; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Graft Occlusion, Vascular
MeSH Terms: conditions — Graft Occlusion, Vascular | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Open aortic repair: 145 patients with open aortic repair for abdominal aortic aneurysmal disease (n=139) or abdominal aortic occlusive disease (n=89)
  Interventions: Procedure: Aortic repair
- Laparoscopic aortic repair: 83 patients with Laparoscopic aortic repair for abdominal aortic aneurysmal disease (n=30) or abdominal aortic occlusive disease (n=53)
  Interventions: Procedure: Aortic repair

INTERVENTIONS:
Procedure: Aortic repair — Aortic bypass

SUMMARY:
This prospective study was designed to analyse the postoperative and long-term outcomes of total laparoscopic vs. open surgical repair of infra-renal abdominal aortic occlusive disease (AOD) and infra-renal aortic aneurysmal disease (AAA) in comparable groups of patients using a propensity analysis model.

DETAILED DESCRIPTION:
From January 2006 to January 2010, 228 consecutive patients who received an aortic bypass for AAA (n=139) or for AOD (n=89) were studied. Open repair was performed in145 patients (AAA=109, AOD=36) and total laparoscopic repair in 83 patients (AAA=30, AOD=53). One-to-one propensity score matching between study groups was done according to a difference in the logit of propensity score of less than 0.04 between each patient pairs in the study groups. Logistic regression with the help of backward selection was used to adjust the effect of treatment method for propensity score as well as other variables in evaluating postoperative and long-term outcome. A p value < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aortic occlusive disease (TASC C & D)
* Aortic abdominal aneurysm with a diameter > 5 cm

Exclusion Criteria:

* Patients with an occlusive disease amenable to stenting (TASC A & B)
* Patients with an abdominal aortic aneurysm with an anatomy allowing the use of a stent graft (EVAR)
* Patients with a life expectancy < 3 years or ASA 4 with a high operative risk

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with an abdominal aortic aneurysm or an occlusive aortic disease operated from January 2006 to January 2010.
  Open repair was performed in145 patients (AAA=109, AOD=36) Total laparoscopic repair was performed in 83 patients (AAA=30, AOD=53).
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Composite adverse events (bypass occlusion, bleeding, graft infection, redo) | 0 to 6 years postoperative
  Any of these complications occurring during this time frame

SECONDARY OUTCOMES:
Mortality | 0 to 6 years postoperative
  Any death occurring within the first 30 days and after

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Ricco, MD, PhD, Principal Investigator — CHU, University of Poitiers, medical school

REFERENCES:
- [Derived] Ricco JB, Cau J, Schneider F, Desvergnes M, Lefort N, Belmonte R. Chirurgie aortique totalement laparoscopique ou par laparotomie: comparaison des resultats apres appariement par un score de propension. Bull Acad Natl Med. 2016 Mar;200(3):527-40; discussion 540-3. French. PMID 28644602
- [Derived] Ricco JB, Cau J, Biancari F, Desvergnes M, Lefort N, Belmonte R, Schneider F. Outcome After Open and Laparoscopic Aortic Surgery in Matched Cohorts Using Propensity Score Matching. Eur J Vasc Endovasc Surg. 2016 Aug;52(2):179-88. doi: 10.1016/j.ejvs.2016.02.021. Epub 2016 Apr 18. PMID 27102201